CLINICAL TRIAL: NCT06604286
Title: Postoperative Dexamethasone Injected Into Masseter Muscle and Pterygomandibular Space After Mandibular Third Molar Surgery; Comparison of Effects on Pain, Edema and Trismus
Brief Title: Comparison of the Effects of Intraoral Postoperative Dexamethasone Applications After Mandibular Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Muhammet Yasin Pektaş, research assistant, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 23.DUS.002
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Wisdom Teeth; Edema Face; Trismus; Pain, Postoperative
Keywords: Dexamethasone; Third Molar Surgery; edema; trismus; Mandibula
MeSH Terms: conditions — Trismus; Pain, Postoperative; Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 8 mg IM dexamethasone injection into the masseter muscle (Active Comparator): Group 1 (Masseter Injection) (n=20): 8 mg IM dexamethasone injection into the masseter muscle of the patients in this group was performed.
  Dexamethasone injection in group 1 was made into the masseter muscle. Injection; The margo anterior of the mandible was palpated and horizontally parallel to the occlusal level of the mandibular second molar tooth and 1 cm behind the margo anterior towards the mandibular ramus. Bone contact was not taken during the injection and the injection was made by taking negative aspiration.Similar to the mandibular anesthesia technique
  Interventions: Drug: In this group, patients received 8 mg IM dexamethasone injection into the masseter muscle after impacted tooth surgery.
- 8 mg IM dexamethasone injection into the pterygomandibular cavity (Active Comparator): Group 2 (Pterygomandibular Space Injection) (n=20): 8 mg IM dexamethasone injection into the pterygomandibular cavity of the patients in this group was performed.
  The injection given to Group 2 was directed to the region between the margo anterior of the mandible and the raphe pterygomandibularis, 1 cm above the occlusal level of the mandibular 2nd molar tooth, and the direction of the syringe from the incisal top of the opposing mandibular canine tooth to this region, and then entering the pterygomandibular cavity. Bone contact was not taken during the injection and the injection was made by taking negative aspiration
  Interventions: Drug: 8 mg IM dexamethasone injection into the pterygoid cavity after impacted tooth surgery.

INTERVENTIONS:
Drug: In this group, patients received 8 mg IM dexamethasone injection into the masseter muscle after impacted tooth surgery. — 8 mg IM dexamethasone injection was given to the groups immediately after the operation area was sutured after impacted dental surgery. Dexamethasone injection in group 1 was made into the masseter muscle. injection; The margo anterior of the mandible was palpated and horizontally parallel to the occlusal level of the mandibular second molar tooth and 1 cm behind the margo anterior towards the mandibular ramus. Bone contact was not taken during the injection and the injection was made by taking negative aspiration.
  Other Names: Group 1 (Masseter Injection)
  Arms: 8 mg IM dexamethasone injection into the masseter muscle
Drug: 8 mg IM dexamethasone injection into the pterygoid cavity after impacted tooth surgery. — 8 mg IM dexamethasone injection was given to the group immediately after the operation area was sutured after impacted dental surgery. Dexamethasone injection given to Group 2 was directed to the region between the margo anterior of the mandible and the raphe pterygomandibularis, 1 cm above the occlusal level of the mandibular 2nd molar tooth, and the direction of the syringe from the incisal top of the opposing mandibular canine tooth to this region, and then entering the pterygomandibular cavity.
  Other Names: Group 2 (Pterygomandibular Space Injection)
  Arms: 8 mg IM dexamethasone injection into the pterygomandibular cavity

SUMMARY:
The aim of this study is to comparatively evaluate the effects of dexamethasone injected into the masseter muscle and pterygomandibular space after mandibular third molar surgery on postoperative pain, edema, trismus and quality of life.

This clinical study will include 20 patients aged 18-25 years who underwent extraction of bilaterally impacted mandibular third molars in 2 consecutive sessions. The patients will randomly divide into two groups; Group 1 (n = 20) received 8 mg IM dexamethasone injection into the masseter muscle after the surgical procedure and Group 2 (n = 20) received 8 mg IM dexamethasone injection into the pterygomandibular space after the surgical procedure. Postoperative pain will record using the VAS scale at 6 hours, 12 hours, 24 hours, 2 and 7 days postoperatively. Edema, salivary cortisol and postoperative oral health quality of life and patient satisfaction will evaluate before surgery and on the 2nd and 7th days after surgery.

DETAILED DESCRIPTION:
Our study aims to reduce pain, edema and restricted mouth opening (trismus) that are frequently seen after impacted tooth extraction operations with steroid applied locally to the area where the operation is performed.

Our aim in this study is to compare the effectiveness of dexamethasone (steroid) applied to different areas in terms of pain, edema and trismus by injecting dexamethasone 8 mg/2 ml into the masseter muscle immediately after the operation in the first operation and dexamethasone 8 mg/2 ml into the pterygomandibular space immediately after the operation in the second (symmetrically impacted tooth) operation in volunteer patients with bilateral and symmetrically impacted lower third molars after tooth extraction surgery.

Conditions for Participation in the Study:

Regardless of gender, over 18 years of age; Volunteer patients with bilateral, symmetrical, bone-retained impacted wisdom teeth in the mandible, Volunteer patients without any systemic disease, Volunteer patients who will voluntarily sign the informed consent form, informed about the duration, purpose and requirements of the study.

Duration of the Study: In the study, your bilateral impacted teeth will be extracted at 2-week intervals. There will be check-ups on the day of the procedure, 3rd and 7th days after both procedures, and the study will last a total of 1 month for a volunteer patient.

Number of Volunteers: The number of volunteers expected to participate in the study is 20.

Treatments to be Applied in the Study: In our study, your 2 impacted mandibular third molars will be extracted and immediately after the procedure; since the area is under anesthesia, steroid medication will be injected around the extraction areas without any pain.

Interventional Methods to be Applied in the Study: In this study, dexamethasone 8mg/2ml, which is recommended as a treatment method to reduce complications after impacted tooth surgery in Oral, Dental and Maxillofacial Surgery clinics and which we routinely use in our clinic in many surgical procedures including especially difficult impacted tooth extractions (complicated tooth extraction, periodontal surgical procedures, sinus elevation, dental implant surgery, and intraoral graft applications, etc.), will be injected into two different areas (masseter muscle and pterygomandibular area) within the operation field and under the effect of anesthesia in a painless and practical way immediately after the operation; and its effects in terms of pain, edema and trismus will be compared. Experimental Parts of the Study: Volunteer patients to be included in the study will be compared with the edema, trismus and pain scale tests of the steroid injected around the operation area on both sides but in different places after the extraction of their impacted teeth at 2-week intervals. Before the procedure, at the 6th hour, 12th hour, 1st day, 2nd day and 7th day follow-ups; Pain Scale (VAS), Oral Health Impact Profile (OHIP-14) questionnaire, before the surgical procedure and at the 6th hour, 12th hour, 1st, 2nd and 7th day post-op saliva samples will be collected and the amount of salivary cortisone at these times will be measured and compared and edema and trismus (limited mouth opening) measurements will be made and evaluated in terms of different parameters and recorded in the follow-ups. Treatment Risks

Allergic reactions, low/high blood pressure and temporary facial paralysis may be observed after local anesthesia, although rare, Allergic reactions to dexamethasone may develop, although rare, Swelling or redness, discomfort in the surgical area, Redness and cracking due to tension in the corners of the mouth, Infection and delayed wound healing, Dry socket; jaw pain that usually starts a few days after surgery due to inadequate care; more common in lower jaw extractions, especially wisdom teeth.

Damage to adjacent teeth, especially in the presence of large fillings and crowns, Loss of sensation or decreased sensation in the gums, lips, tongue, teeth and tip of the jaw. It can be seen especially in teeth with roots close to the nerves, such as wisdom teeth. Numbness almost always returns to normal, but very rarely can be permanent.

Trismus; limitation of mouth opening due to inflammation or swelling. Most surgical procedures are routine and no major complications are expected. Complications that do occur are minor and easily treatable. What are your responsibilities? During the study, you must follow your doctor recommendations after the procedure and come to follow-up appointments on the 3rd and 7th days. If you encounter any problems during the study, you must notify your doctor.

Participation in this study is entirely voluntary. You can refuse to take part in the study or withdraw from the study at any stage; even in the event of refusal or withdrawal, your subsequent treatment process will be guaranteed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with no systemic disease, AAD (American Society of Anesthesiologists) class I and BMI (body mass index) below 30.

  2. Patients between the ages of 18-25 with bilaterally symmetrical and mesioangularly positioned impacted third molars in the mandible.

  3. Patients with impacted mandibular third molars in class II-B according to the Pell and Gregory classification.

  4. Patients with impacted third molars that are fully or partially retained and asymptomatic.

  5. Patients with impacted mandibular third molars that are not associated with any pathology such as cysts or tumors and do not have active perichronitis.

  6. Patients with at least 2/3 of root development completed.

  7. Patients without complaints such as active caries, periodontal disease, pain or swelling in the operation area.

  8. Patients without a history of infection or perichronitis in the operation area.

Exclusion Criteria:

* 1. Patients with a history of allergy to dexamethasone or other drugs to be used in the study.

  2. Patients with systemic bacterial, viral, and fungal infections.

  3. Breastfeeding mothers.

  4. Patients with diagnosed or suspected pregnancies.

  5. Patients in whom corticosteroids are contraindicated.

  6. Patients who have recently been treated with anti-inflammatory drugs.

  7. Patients with cardiovascular disease.

  8. Patients with acute or chronic maxillary sinusitis.

  9. Patients who are taking medications such as antidepressants or antihistamines on a regular basis.

  10. Patients with psychiatric problems.

  11. Patients with diabetes mellitus, rheumatic diseases, hematological diseases, or liver diseases.

  12. Patients at risk of effective endocarditis.

  13. Patients who smoke.

  14. Patients who use oral contraceptives.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-04-27 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain | Patients were called for control at the 6th, 12th, 24th hour, 2nd and 7th days postoperatively, and the forms were filled out verbatim by the researcher.
  In order to ensure standardization in the use of analgesic drugs, all patients; It was explained in writing and verbally that he should take the first medicine 1 hour after the end of the operation, and that if he had pain in the future, he could take analgesic medicine 3 times a day, one every 8 hours. The use of analgesic medication other than the specified analgesic use by the patients during the 1-week period after the surgical procedure was recorded. Pain assessment was made using VAS scales numbered from 0 to 10.
Evaluation of Edema | preoperative and postoperative days 2-7
  In postoperative edema evaluation; The distances between some anatomical points on the face were measured on preoperative and postoperative days 2-7 and the changes between these lengths were calculated. The tragus, soft tissue pogonion, lateral canthus of the eye, gonion point in the mandibular angle and commissure labiorum were used as anatomical reference points. In measurements; The patient was seated upright and the lengths of tragus-lateral canthus, tragus-commissura loborum, tragus-soft tissue pogonion, tragus-gonion and gonion-lateral canthus were measured with a flexible ruler and calculated linearly
Evaluation of Trismus | preoperative and postoperative days 2-7
  Trismus; It was evaluated using the measurement of the distances between the mesial corners of the incisal edge of the left maxillary and mandibular central teeth at maximum mouth opening, on preoperative and postoperative days 2-7.
Evaluation of Salivary Cortisol Amount | preoperative and postoperative days 2-7
  Saliva samples were collected from the patients immediately before the surgical procedures and on postoperative days 2 and 7. Salivary cortisol ELISA kits (ELK Biotechnology ELK8526 Human Cor(Cortisol) ELISA Kit) with a sensitivity of 1.02 ng/mL and a detection range of 3.13-200 ng/mL were used to analyze salivary cortisol.
Evaluation of Oral Health Related Quality of Life and Patient Satisfaction After Surgery | preoperative and postoperative days 2-7
  The OHIP-14 form was used to assess oral health-related quality of life and patient satisfaction after the surgical procedure on preoperative and postoperative days 2-7. The OHIP-14 form was used to assess seven main categories: functional limitations, physical pain, psychological discomfort, physical disability, social disability, psychological disability and handicap. In addition, the total OHIP-14 score was calculated and evaluated by summing the scores given to all questions of the oral health impact profile form.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Yasin Pektaş, Principal Investigator — Afyonkarahisar Health Science University
Locations (1):
- Afyonkarahisar Health Sciences University Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Afyonkarahisar, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vivek GK, Vaibhav N, Shetty A, Mohammad I, Ahmed N, Umeshappa H. Efficacy of Various Routes of Dexamethasone Administration in Reducing Postoperative Sequelae Following Impacted Third Molar Surgery. Ann Maxillofac Surg. 2020 Jan-Jun;10(1):61-65. doi: 10.4103/ams.ams_66_19. Epub 2020 Jun 8. PMID 32855917
- [Background] Chaudhary PD, Rastogi S, Gupta P, Niranjanaprasad Indra B, Thomas R, Choudhury R. Pre-emptive effect of dexamethasone injection and consumption on post-operative swelling, pain, and trismus after third molar surgery. A prospective, double blind and randomized study. J Oral Biol Craniofac Res. 2015 Jan-Apr;5(1):21-7. doi: 10.1016/j.jobcr.2015.02.001. Epub 2015 Mar 5. PMID 25853044
- [Background] Bhargava D, Sreekumar K, Deshpande A. Effects of intra-space injection of Twin mix versus intraoral-submucosal, intramuscular, intravenous and per-oral administration of dexamethasone on post-operative sequelae after mandibular impacted third molar surgery: a preliminary clinical comparative study. Oral Maxillofac Surg. 2014 Sep;18(3):293-6. doi: 10.1007/s10006-013-0412-7. Epub 2013 Mar 20. PMID 23512235
- [Background] Antunes AA, Avelar RL, Martins Neto EC, Frota R, Dias E. Effect of two routes of administration of dexamethasone on pain, edema, and trismus in impacted lower third molar surgery. Oral Maxillofac Surg. 2011 Dec;15(4):217-23. doi: 10.1007/s10006-011-0290-9. Epub 2011 Aug 16. PMID 21845387